CLINICAL TRIAL: NCT04327817
Title: A Prospective Single Arm Pilot Study to Investigate the Dynamic Brain and Multifidus Muscle Imaging in Response to Multifidus Stimulation in Patients With Low Back Pain Undergoing Reactiv8 Implant
Brief Title: Multifidus PET Scan Study
Acronym: MUST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Mainstay Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 254110
Record Dates: First submitted 2020-03-27; First posted 2020-03-31 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Low Back Pain
Keywords: Multifidus stimulation; 18F FDG PET/CT scans; Multifidus muscle
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: The Mainstay ReActiv8 is an implantable electrical stimulation system that consists of an implantable pulse generator, implantable leads, programmer, activator and magnet.
Masking Description: The ReActiv8 IPG, and the ReActiv8 leads (available in either 45 cm or 65 cm lengths), plus suture sleeves.
  The Lead is designed to be placed using a commercially available 7 Fr Introducer Kit (not included with ReActiv8) and the Mainstay Model TUN1 Tunneler (included with ReActiv8) or commercially available equivalent. The electrodes are located at the distal end of a Stimulation Lead that is connected to an implantable pulse generator (IPG) placed in a surgical pocket typically above the buttocks (in a place similar to that used in Spinal Cord Stimulation implants). Two leads are placed (one each left and right side) and connected to the IPG. The IPG is externally programmable with a Programmer. Stimulation is manually initiated by an external device (Activator) and can be stopped with the Activator or Magnet.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Multifidus ReActiv8 stimulator (Other): The Mainstay ReActiv8 is an implantable electrical stimulation system that consists of an implantable pulse generator, implantable leads, programmer, activator and magnet.
  Interventions: Device: Multifidus stimulator

INTERVENTIONS:
Device: Multifidus stimulator — Patient eligible for the study and have provided consent will have a baseline PET scan. Multifidus ReActiv8 Stimulator will be inserted using standard treatment for lumbar pain at Barts Health NHS Hospitals.
  All patients who receive the Reactiv8 system will continue to receive multifidus stimulation 20Hz for the next 6 months as per standard of care of multifidus stimulation; at the end of this period, the patients will undergo PET scanning and questionnaires. Thereafter, stimulation will continue and 3rd PET scan will be performed at 1year post implant.
  Other Names: ReActiv8 stimulator

SUMMARY:
The study involves investigating phenotypic changes (ie metabolic activity in brain pain matrix areas, metabolic activity and textural analysis of multifidus muscle) following multifidus stimulation and establishing relationship with the change in pain, functionality and quality of life.

DETAILED DESCRIPTION:
Multifidus Stimulation via the dorsal ramus is an effective therapy for patients with intractable low back pain. Barts Health has had a positive experience following the implantation of Reactiv8 stimulator in patients with very good success rate in both in Reactiv8 A & B studies. Multifidus stimulation (MS) serves an advantage of functional restoration and neuro-rehabilitation in this difficult group of patients of intractable low back pain, however objective measurement of the multifidus stimulation on supraspinal pathways particularly the changes in higher centres in the brain and in the multifidus muscle itself remains to be characterised.

Dynamic brain imaging in pain (PET/CT scans) Dynamic brain imaging is increasingly used as a research tool to understand the mechanisms of pain and also pain interventions. This is done by using either a functional MRI (fMRI) or Positron Emission Tomography (PET-CT). The implant used for stimulation of the multifidus muscle is not MRI compatible which precludes the use of fMRI. Hence PET-CT is the best available option to investigate the changes in the brain in patients having MS. Functional changes in the brain are identified by the changes in the regional cerebral blood flow (rCBF) as determined by the changes in the distribution of the radioactiove contrast F18- fluorodeoxyglucose (18-FDG) in different areas of the brain.

PET/CT in chronic pain: Chronic pain has been associated with changes in brain structure as well as metabolism especially in the second somatic (SII) regions, insula and anterior cingulate cortex (ACC). Less consistently, changes have also been seen in thalamus and primary somatic area (SI). Sensory discrimination, summation, affect, cognition and attention all seem to influence different areas of the brain there by modulate the patient's pain perception. There is some evidence to suggest that some of these changes may be altered with treatment using either medications or other interventions.

PET in spinal cord stimulation (SCS): There is limited data available on functional neuroimaging following SCS. Nishai et al. conducted FDG PET Scanning in 20 patients (7 CRPS and 13 control) and reported increase in FDG (Flurodeoxyglucose) uptake in left thalamus, anterior cingulate cortex, bilateral insula, dorsolateral prefrontal cortex and bilateral temporal gyrus in six patients where SCS is effective. Similarly Kishima et al reported an increase in blood fIow following SCS in thalamus, orbitofrontal, parietal and prefrontal cortex proportional to the pain relief (larger PET assessed increase in rCBF correlates with decrease in pain intensity) It has been postulated that thalamus activity may relate to whether SCS is effective or not. Recent study comparing Tonic Vs Burst frequencies established differential brain pain matrix areas stimulation with PET-FDG demonstrating the fact of Burst being more associated with medial pathway stimulation, hence perception.

PET in Dorsal Root Ganglion (DRG) stimulation: Barts Health presented the first data on L2-DRG stimulation for low back pain in virgin back patients, with identifiable changes in cereberal metabolic activity in insula, PAG, cerebral cortex following L2-DRG stimulation. Metabolic activity at the target area was measured as standardized uptake value and response to individual pain matrix were demonstrated following L2 stimulation. SUVmax (maximum standardised uptake value) is one of the most common way to measure glucose metabolism. There is evidence that in patients with brain tumours there is increase in cerebral glucose metabolism (measured with SUVmax before and after cervical spinal cord stimulation).

Textural Analysis: Tissue heterogeneity is an important feature associated with adverse tissue biology. Textural analysis has been validated an emerging technique for assessing tissue heterogeneity and quantitative assessments of tissue heterogeneity has the potential to provide non-invasive imaging biomarkers of prognosis and treatment response. Clinical studies have indicated the ability of CT texture analysis (CTTA) to provide independent predictors of survival for patients with malignancies and marker of treatment response. We are utilising the same principal using low dose CT which will be acquired as part of 18F FDG PET-CT image examination. There is no additional radiation exposure for textural analysis. The filtration-histogram method comprises an initial filtration step that highlights image features of a specific size, followed by histogram analysis of the filtered image. The standard descriptors include mean, standard deviation, skewness and kurtosis.

There is still limited data on brain imaging within neuromodulation and there is currently no looking at the PET-CT scan changes following multifidus stimulation. Hence this would be the first study looking into the dynamic brain imaging changes following multifidus stimulation.

This study aims to investigate the dynamic brain imaging in pain using PET scan in patients who have undergone successful Reactiv8 implantation. This may provide us with information on the nature of changes occurring in the brain following multifidus stimulation in the brain pain matrix. Additionally, we aim to measure the changes in the multifidus consistency and metabolic activity following stimulation. This will also hopefully enable us to correlate it with the changes in clinical and health related outcome questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥22 years, ≤75 years
2. Low Back Pain VAS of ≥6.0cm and ≤9.0cm (on a 10cm scale) at the Baseline Visit.
3. Oswestry Disability Index score ≥21% and ≤60% at the Baseline Visit
4. Chronic Low Back Pain defined as pain and discomfort localized below the costal margin and above the inferior gluteal fold (with or without referred leg pain) that has persisted >90 days prior to the Baseline Visit, which has resulted in pain in at least half of the days in the 12 months prior to the Baseline Visit, as reported by the Subject.
5. Evidence of lumbar multifidus muscle dysfunction (for example by the Prone Instability Test (PIT)).
6. Continuing low back pain despite >90 days of medical management including:

   1. At least one attempt of physical therapy treatment for low back pain, which may optionally be accomplished over multiple episodes or flare-ups of low back pain.
   2. For Subjects with medications prescribed and used for chronic low back pain, usage shall be at a stable dose in the 30 days prior to the Baseline Visit as reported by the Subject.

   NOTE: A stable dose means the Subject reports no significant change in regular use of medications, which may include PRN use, in the 30 days prior to the Baseline Visit. Typical use must be provided
7. Be willing and capable of giving Informed Consent.
8. Ability to comply with the instructions for use and to operate ReActiv8, and to comply with this Clinical Investigation Plan.
9. Suitable for ReActiv8 surgery as determined by the implanting physician prior to inclusion.

Exclusion Criteria:

1. BMI > 35
2. Back Pain characteristics:

   1. Any surgical correction procedure for scoliosis at any time, or a current clinical diagnosis of moderate to severe scoliosis (Cobb angle ≥25°).
   2. Lumbar spine stenosis, as defined by an anterior-posterior diameter of the spinal canal <10mm in Subjects with lower extremity pain.
   3. Neurological deficit possibly associated with the back pain (e.g. foot drop).
   4. Back pain due to pelvic or visceral reasons (e.g.: endometriosis or fibroids) or infection (e.g.: post herpetic neuralgia).
   5. Back pain due to inflammation or damage to the spinal cord or adjacent structures (e.g. arachnoiditis or syringomyelia).
   6. Pathology seen on MRI that is clearly identified and is likely the cause of the CLBP that is amenable to surgery.
   7. Back pain due to vascular causes such as aortic aneurysm and dissection.
3. Leg pain described as being worse than back pain, or radiculopathy (neuropathic pain) below the knee.
4. Source of pain is the sacroiliac joint as determined by the Investigator.
5. Drug use per Subject report as follows:

   a. Current baseline use of >120mg oral morphine equivalent per day of opioids. b. Current use of breakthrough dose of >60mg oral morphine equivalent per day. c. Current requirement of opioids for treatment of a condition other than low back pain.

   d. History of any substance abuse at any time in the five years prior to the Baseline Visit.

   e. Currently taking >15mg Diazepam per day or equivalent.
6. Surgical or other procedures exclusions:

   1. Any previous rhizotomy or rhizolysis procedure, including cryoablation, RF ablation or pulsed RF on the dorsal root ganglion (DRG) or the medial branch of the dorsal ramus nerve that crosses or lies below the T8 vertebra, within one year prior to the Baseline Visit.
   2. Anesthetic block of the DRG or medial branch of dorsal ramus nerve that crosses or lies below the T8 vertebra or injection of epidural steroids for back pain in the 30 days prior to the Baseline Visit.
   3. Any previous back surgery including laminectomy or discectomy at or below segmental level T8, or spinal fusion at any level.
   4. Any previous thoracic or lumbar sympathectomy.

8. Any prior diagnosis of lumbar vertebral compression fracture, lumbar pars fracture, pars defect, or lumbar annular tear with disc protrusion that is amenable to surgery.

9 Any co-morbid chronic pain conditions. 10. Other clinical conditions:

1. Pregnant or planning to be pregnant in the next 24 months, at the time of inclusion.
2. Pregnancy at any time in the 6 months, or lactating at any time in the 3 months, prior to the Baseline Visit.
3. Any condition unrelated to the CLBP such as muscle wasting, muscle atrophy, other disability (e.g.: paraplegic, amputee, cerebral palsy) or muscular or skeletal disease (e.g.: arthritis in trunk or limbs, multiple sclerosis, rheumatoid arthritis) which, in the opinion of the Investigator, could limit physical movement or compliance with the protocol, or interfere with the assessment of efficacy of the investigational procedure.
4. Poorly controlled diabetes (Type I or Type II) determined by HbA1c >8.
5. Past or current neurological disorders (e.g.: known multiple sclerosis, motor neuron disease, Guillain-Barré syndrome, Parkinson's, Huntington's Disease, Alzheimer's, epilepsy, stroke, brain cancer, traumatic brain injury).
6. Cancer requiring treatment during the study.
7. Any drugs (e.g.: immunosuppressive drugs) or co-morbidity that might inhibit wound healing or electrode scarring, or drugs associated with reduced effectiveness of neuromodulation for other applications.
8. Any medical condition requiring anticoagulation (other than aspirin) that, in the opinion of the physician prescribing the anticoagulant, cannot be safely suspended for 5 days prior to device implantation surgery and an appropriate period after implantation surgery.
9. Any active infection in the vicinity of the implant site or any systemic infection.

   11. Psycho-social exclusions:

a. Be involved in an injury claim under current litigation. b. Have a pending or approved financial compensation claim (e.g., worker's compensation claim, long term disability claims) or any financial compensation (including social welfare payments) related to the Subject's CLBP.

c. Current incarceration (prison or jail) d. Have an assessment of current active depression significant enough (DASS depression score >18 to impact perception of pain, compliance with intervention and/or ability to evaluate treatment outcome.

e. Have evidence of an active disruptive psychological or psychiatric disorder or other known condition significant enough to impact perception of pain, compliance with intervention and/or ability to evaluate treatment outcome (e.g.: active depression, bipolar disease, Alzheimer's disease) as determined by a psychologist or psychiatrist during the multidisciplinary team meeting to assess suitability of patients.

13. Protocol Compliance Exclusions:

a. Inability or unwillingness to comply with all protocol requirements. b. Inability to maintain the prone or side lying position in a relaxed manner for the duration of each stimulation session.

c. Inability to operate the Activator, such as arthritis that limits arm or shoulder movement, or inability to learn how to operate.

d. Inability to assess changes in pain intensity or perform wound care. e. Inability or unwillingness to complete the Pain score diary. 14. General exclusions:

1. Any other active implantable device including an implantable device for back pain (such as an implantable drug pump or Spinal Cord Stimulator), pacemaker, implantable defibrillator, cochlear implant, deep brain stimulator, or other implanted neurostimulation device.
2. Prior exposure to an implantable neurostimulator for treatment of pain, including spinal cord stimulation (including trial implant of SCS leads), occipital nerve stimulation or peripheral nerve stimulation.
3. A condition currently requiring or likely to require use of MRI or diathermy while implanted with the ReActiv8.
4. Therapy with any investigational intervention (drugs, devices, or procedures) for the treatment of back pain at the time of the Baseline Visit, or at any time in the past if the past investigational intervention did not subsequently gain regulatory approval.
5. Current or planned participation in any clinical trial during participation in this Trial.
6. Life expectancy <1 year.

Ages: 22 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-17 (Actual)

PRIMARY OUTCOMES:
Low Back Pain Visual Analog Scale (VAS) | Baseline
  The instrument used for evaluating pain is the continuous Visual Analog Scale comprised of a horizontal line 10cm in length, anchored by 2 verbal descriptors. The scoring of the scale 0 represents no pain and 10 being the worst pain imaginable.
Low Back Pain Visual Analog Scale (VAS) | 3 months
  The instrument used for evaluating pain is the continuous Visual Analog Scale comprised of a horizontal line 10cm in length, anchored by 2 verbal descriptors. The scoring of the scale 0 represents no pain and 10 being the worst pain imaginable.
Low Back Pain Visual Analog Scale (VAS) | 6 months
  The instrument used for evaluating pain is the continuous Visual Analog Scale comprised of a horizontal line 10cm in length, anchored by 2 verbal descriptors. The scoring of the scale 0 represents no pain and 10 being the worst pain imaginable.
Low Back Pain Visual Analog Scale (VAS) | 12 months
  The instrument used for evaluating pain is the continuous Visual Analog Scale comprised of a horizontal line 10cm in length, anchored by 2 verbal descriptors. The scoring of the scale 0 represents no pain and 10 being the worst pain imaginable.
Low Back Pain Visual Analog Scale (VAS) | 24 months
  The instrument used for evaluating pain is the continuous Visual Analog Scale comprised of a horizontal line 10cm in length, anchored by 2 verbal descriptors. The scoring of the scale 0 represents no pain and 10 being the worst pain imaginable.
Oswestry Disability Index (ODI) | Baseline
  Oswestry Disability Index (ODI) is a disease specific assessment of the disabling effects of back pain. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability.
Oswestry Disability Index (ODI) | 3 months
  Oswestry Disability Index (ODI) is a disease specific assessment of the disabling effects of back pain. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability.
Oswestry Disability Index (ODI) | 6 months
  Oswestry Disability Index (ODI) is a disease specific assessment of the disabling effects of back pain. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability.
Oswestry Disability Index (ODI) | 12 months
  Oswestry Disability Index (ODI) is a disease specific assessment of the disabling effects of back pain. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability.
Oswestry Disability Index (ODI) | 24 months
  Oswestry Disability Index (ODI) is a disease specific assessment of the disabling effects of back pain. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability.
European Quality of Life Score on Five Dimensions (EQ-5D) | Baseline
  The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The answers given to ED-5D can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health.
European Quality of Life Score on Five Dimensions (EQ-5D) | 3 months
  The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The answers given to ED-5D can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health.
European Quality of Life Score on Five Dimensions (EQ-5D) | 6 months
  The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The answers given to ED-5D can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health.
European Quality of Life Score on Five Dimensions (EQ-5D) | 12 months
  The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The answers given to ED-5D can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health.
European Quality of Life Score on Five Dimensions (EQ-5D) | 24 months
  The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. The answers given to ED-5D can be converted into EQ-5D index an utility scores anchored at 0 for death and 1 for perfect health.
Clinical Global Impression of change | 3 months
  Clinical Global Impression - Global Improvement consists of a question comparing the subject's situation at baseline to that at each follow-up visit and it to be completed by the Investigator. A 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. 1 being very much improved to 7 very much worse.
Clinical Global Impression of change | 6 months
  Clinical Global Impression - Global Improvement consists of a question comparing the subject's situation at baseline to that at each follow-up visit and it to be completed by the Investigator. A 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. 1 being very much improved to 7 very much worse.
Clinical Global Impression of change | 12 months
  Clinical Global Impression - Global Improvement consists of a question comparing the subject's situation at baseline to that at each follow-up visit and it to be completed by the Investigator. A 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. 1 being very much improved to 7 very much worse.
Clinical Global Impression of change | 24 months
  Clinical Global Impression - Global Improvement consists of a question comparing the subject's situation at baseline to that at each follow-up visit and it to be completed by the Investigator.
Pain and Sleep 3 point index (PSQ-3) | Baseline
  The PSQ-3 is an instrument that measures the quality of sleep over a month. This questionnaire is based on 3 questions about sleep and marked as 10cm visual scale where 0 is no problem sleeping to 10 being always having trouble sleeping.
Pain and Sleep 3 point index (PSQ-3) | 3 months
  The PSQ-3 is an instrument that measures the quality of sleep over a month. This questionnaire is based on 3 questions about sleep and marked as 10cm visual scale where 0 is no problem sleeping to 10 being always having trouble sleeping.
Pain and Sleep 3 point index (PSQ-3) | 6 months
  The PSQ-3 is an instrument that measures the quality of sleep over a month. This questionnaire is based on 3 questions about sleep and marked as 10cm visual scale where 0 is no problem sleeping to 10 being always having trouble sleeping.
Pain and Sleep 3 point index (PSQ-3) | 12 months
  The PSQ-3 is an instrument that measures the quality of sleep over a month. This questionnaire is based on 3 questions about sleep and marked as 10cm visual scale where 0 is no problem sleeping to 10 being always having trouble sleeping.
Pain and Sleep 3 point index (PSQ-3) | 24 months
  The PSQ-3 is an instrument that measures the quality of sleep over a month. This questionnaire is based on 3 questions about sleep and marked as 10cm visual scale where 0 is no problem sleeping to 10 being always having trouble sleeping.
PainDETECT Questionnaire | baseline
  The PainDETECT questionnaire (PD-Q) is a screening tool specifically designed to identify neuropathic pain in an heterogenous low back pain cohort.Scores on the nine-item painDETECT (seven pain-symptom items, one pain-course item, one pain-irradiation item) range from -1 to 38 (worst Neuropathic pain); the seven-item painDETECT scores (only pain symptoms) range from 0 to 35.
PainDETECT Questionnaire | 3 months
  The PainDETECT questionnaire (PD-Q) is a screening tool specifically designed to identify neuropathic pain in an heterogenous low back pain cohort.Scores on the nine-item painDETECT (seven pain-symptom items, one pain-course item, one pain-irradiation item) range from -1 to 38 (worst Neuropathic pain); the seven-item painDETECT scores (only pain symptoms) range from 0 to 35.
PainDETECT Questionnaire | 6 months
  The PainDETECT questionnaire (PD-Q) is a screening tool specifically designed to identify neuropathic pain in an heterogenous low back pain cohort.Scores on the nine-item painDETECT (seven pain-symptom items, one pain-course item, one pain-irradiation item) range from -1 to 38 (worst Neuropathic pain); the seven-item painDETECT scores (only pain symptoms) range from 0 to 35.
PainDETECT Questionnaire | 12 months
  The PainDETECT questionnaire (PD-Q) is a screening tool specifically designed to identify neuropathic pain in an heterogenous low back pain cohort.Scores on the nine-item painDETECT (seven pain-symptom items, one pain-course item, one pain-irradiation item) range from -1 to 38 (worst Neuropathic pain); the seven-item painDETECT scores (only pain symptoms) range from 0 to 35.
PainDETECT Questionnaire | 24 months
  The PainDETECT questionnaire (PD-Q) is a screening tool specifically designed to identify neuropathic pain in an heterogenous low back pain cohort.Scores on the nine-item painDETECT (seven pain-symptom items, one pain-course item, one pain-irradiation item) range from -1 to 38 (worst Neuropathic pain); the seven-item painDETECT scores (only pain symptoms) range from 0 to 35.
Percent Pain Relief | 3 months
  the Subject is asked to report the percent pain relief at the time of the current visit compared to the pain at baseline. The scale is marked at 0% with no change to 100% total change.
Percent Pain Relief | 6 months
  the Subject is asked to report the percent pain relief at the time of the current visit compared to the pain at baseline. The scale is marked at 0% with no change to 100% total change.
Percent Pain Relief | 12 months
  the Subject is asked to report the percent pain relief at the time of the current visit compared to the pain at baseline. The scale is marked at 0% with no change to 100% total change.
Percent Pain Relief | 24 months
  the Subject is asked to report the percent pain relief at the time of the current visit compared to the pain at baseline. The scale is marked at 0% with no change to 100% total change.
Subject Global Impression of Change (SGIC) | 3 months
  the Subject's overall status since baseline. A 7-point scale that requires the patient to rate the severity of their illness at the time of assessment, relative to the patients's diagnosis.
Subject Global Impression of Change (SGIC) | 6 months
  the Subject's overall status since baseline. A 7-point scale that requires the patient to rate the severity of their illness at the time of assessment, relative to the patients's diagnosis.
Subject Global Impression of Change (SGIC) | 12 months
  the Subject's overall status since baseline. A 7-point scale that requires the patient to rate the severity of their illness at the time of assessment, relative to the patients's diagnosis.
Subject Global Impression of Change (SGIC) | 24 months
  the Subject's overall status since baseline. A 7-point scale that requires the patient to rate the severity of their illness at the time of assessment, relative to the patients's diagnosis.

OTHER OUTCOMES:
PET/CT scans | Baseline
  18F-FDG Positron Emission Tomography/Computed Tomography (PET-CT) assessments will be carried out during this study.
PET/CT scans | 6 months
  18F-FDG Positron Emission Tomography/Computed Tomography (PET-CT) assessments will be carried out during this study.
PET/CT scans | 12 months
  18F-FDG Positron Emission Tomography/Computed Tomography (PET-CT) assessments will be carried out during this study.

CONTACTS AND LOCATIONS:
Overall Officials: Vivek H Mehta, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- Barts Health NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We will follow the policies laid by the local information governance team at Barts Health NHS Trust and NHS code of Confidentiality in accordance to the data protection act.